CLINICAL TRIAL: NCT04274777
Title: The Relationship Between Lipid Peroxidation Products From Traumatic Brain Injury and Secondary Coagulation Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDSJWKTBIC
Record Dates: First submitted 2019-09-24; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2019-10

CONDITIONS: Traumatic Brain Injury; Coagulation Disorder
Keywords: Traumatic Brain Injury; Coagulation Disorder; Lipid Peroxidation
MeSH Terms: conditions — Brain Injuries, Traumatic; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to observe the relationship between the level of lipid peroxidation products in serum of patients with traumatic brain injury and secondary coagulation disorders.

DETAILED DESCRIPTION:
Uncontrolled hemorrhage after trauma is the leading cause of death. The mechanism of secondary coagulation dysfunction after trauma is special and complex, which has not been fully explained, leading to limited treatment and prevention methods. Coagulation disorders caused by traumatic brain injury is a systemic manifestation of local injury, which can activate platelets and promote platelet aggregation, activate thrombin, and promote the production of fibrin, leading to the formation of thrombosis. However, in non-injured areas, pro-coagulant molecules from damaged brain tissue reach the body through the broken blood-brain barrier, and also activate platelets and thrombin, promoting the formation of blood clots. Lipid peroxidation products are closely related to the occurrence of coagulation dysfunction. The effects lipid peroxidation products on platelets, thrombin and anticoagulant pathways may be a novel mechanism of secondary coagulation dysfunction in traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

1. The interval between injury and admission is less than 24 hours
2. Age>18yrs and age<80yrs
3. Non-head abbreviated injury score < 3
4. Did not undertake treatment before enrollment
5. Informed consent to participate in the study

Exclusion Criteria:

1. Take anticoagulants or antiplatelet drugs
2. Smoking history
3. Hemorrhagic or ischemic cerebrovascular disease occurred within six months
4. Other systemic diseases: uremia, cirrhosis, malignant tumor, etc
5. Patients with severe mental illness who are unable to communicate when diagnosed
6. Patients who refused follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All of the traumatic brain injury patients receiving treatment in Tangdu Hospital during 2019-2020
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-21 (Actual); Primary Completion 2020-09-21 (Estimated); Study Completion 2020-12-21 (Estimated)

PRIMARY OUTCOMES:
The level of lipid peroxidation products in subjects' serum | within 24 hours of trauma
  the level of high and low
Coagulation Disorders | within 24 hours of trauma
  aPTT>40s or INR>1.4 or <100 platelets per L

SECONDARY OUTCOMES:
The 24-hour and 3-month Glasgow outcome score (GOS) | from onset to three months

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qu, M.D, Ph.D, Study Chair — Tang-Du Hospital; Shunnan Ge, M.D, Ph.D, Study Director — Tang-Du Hospital; Wenxing Cui, M.D, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tandu Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harhangi BS, Kompanje EJ, Leebeek FW, Maas AI. Coagulation disorders after traumatic brain injury. Acta Neurochir (Wien). 2008 Feb;150(2):165-75; discussion 175. doi: 10.1007/s00701-007-1475-8. Epub 2008 Jan 2. PMID 18166989
- [Background] Epstein DS, Mitra B, O'Reilly G, Rosenfeld JV, Cameron PA. Acute traumatic coagulopathy in the setting of isolated traumatic brain injury: a systematic review and meta-analysis. Injury. 2014 May;45(5):819-24. doi: 10.1016/j.injury.2014.01.011. Epub 2014 Jan 19. PMID 24529718
- [Background] Zehtabchi S, Soghoian S, Liu Y, Carmody K, Shah L, Whittaker B, Sinert R. The association of coagulopathy and traumatic brain injury in patients with isolated head injury. Resuscitation. 2008 Jan;76(1):52-6. doi: 10.1016/j.resuscitation.2007.06.024. Epub 2007 Aug 15. PMID 17706857
- [Background] Maeda T, Katayama Y, Kawamata T, Aoyama N, Mori T. Hemodynamic depression and microthrombosis in the peripheral areas of cortical contusion in the rat: role of platelet activating factor. Acta Neurochir Suppl. 1997;70:102-5. doi: 10.1007/978-3-7091-6837-0_32. PMID 9416292
- [Background] Zhang J, Zhang F, Dong JF. Coagulopathy induced by traumatic brain injury: systemic manifestation of a localized injury. Blood. 2018 May 3;131(18):2001-2006. doi: 10.1182/blood-2017-11-784108. Epub 2018 Mar 5. PMID 29507078
- [Background] Zhao Z, Wang M, Tian Y, Hilton T, Salsbery B, Zhou EZ, Wu X, Thiagarajan P, Boilard E, Li M, Zhang J, Dong JF. Cardiolipin-mediated procoagulant activity of mitochondria contributes to traumatic brain injury-associated coagulopathy in mice. Blood. 2016 Jun 2;127(22):2763-72. doi: 10.1182/blood-2015-12-688838. Epub 2016 Mar 21. PMID 27002118
- [Background] Wu Y, Liu W, Zhou Y, Hilton T, Zhao Z, Liu W, Wang M, Yeon J, Houck K, Thiagarajan P, Zhang F, Shi FD, Wu X, Li M, Dong JF, Zhang J. von Willebrand factor enhances microvesicle-induced vascular leakage and coagulopathy in mice with traumatic brain injury. Blood. 2018 Sep 6;132(10):1075-1084. doi: 10.1182/blood-2018-03-841932. Epub 2018 Jun 25. PMID 29941674
- [Background] Tian Y, Salsbery B, Wang M, Yuan H, Yang J, Zhao Z, Wu X, Zhang Y, Konkle BA, Thiagarajan P, Li M, Zhang J, Dong JF. Brain-derived microparticles induce systemic coagulation in a murine model of traumatic brain injury. Blood. 2015 Mar 26;125(13):2151-9. doi: 10.1182/blood-2014-09-598805. Epub 2015 Jan 27. PMID 25628471
- [Background] Zhou Y, Cai W, Zhao Z, Hilton T, Wang M, Yeon J, Liu W, Zhang F, Shi FD, Wu X, Thiagarajan P, Li M, Zhang J, Dong JF. Lactadherin promotes microvesicle clearance to prevent coagulopathy and improves survival of severe TBI mice. Blood. 2018 Feb 1;131(5):563-572. doi: 10.1182/blood-2017-08-801738. Epub 2017 Nov 21. PMID 29162596
- [Background] Rossaint R, Bouillon B, Cerny V, Coats TJ, Duranteau J, Fernandez-Mondejar E, Filipescu D, Hunt BJ, Komadina R, Nardi G, Neugebauer EA, Ozier Y, Riddez L, Schultz A, Vincent JL, Spahn DR. The European guideline on management of major bleeding and coagulopathy following trauma: fourth edition. Crit Care. 2016 Apr 12;20:100. doi: 10.1186/s13054-016-1265-x. PMID 27072503
- [Background] Hyder AA, Wunderlich CA, Puvanachandra P, Gururaj G, Kobusingye OC. The impact of traumatic brain injuries: a global perspective. NeuroRehabilitation. 2007;22(5):341-53. PMID 18162698
- [Background] Sun Y, Wang J, Wu X, Xi C, Gai Y, Liu H, Yuan Q, Wang E, Gao L, Hu J, Zhou L. Validating the incidence of coagulopathy and disseminated intravascular coagulation in patients with traumatic brain injury--analysis of 242 cases. Br J Neurosurg. 2011 Jun;25(3):363-8. doi: 10.3109/02688697.2011.552650. Epub 2011 Feb 28. PMID 21355766